CLINICAL TRIAL: NCT03855176
Title: Effectiveness of Booster Vaccination With 1 or 2 Doses of Hepatitis A Vaccine Among HIV-infected Patients During an Ongoing Outbreak in Taiwan
Brief Title: Effectiveness of Booster With 1 or 2 Doses of HAV Vaccine Among HIV-infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201608071MINB
Record Dates: First submitted 2017-09-12; First posted 2019-02-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Hepatitis A; Human Immunodeficiency Virus; Vaccine Response Impaired
MeSH Terms: conditions — Hepatitis A; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1-dose group (Active Comparator): Provide 1 booster dose of HAV vaccine (Vaqta Injectable Product) to those who failed to response after primary HAV vaccination.
  Interventions: Drug: Vaqta Injectable Product
- 2-dose group (Experimental): Provide 2 booster doses of HAV vaccine (Vaqta Injectable Product) to those who failed to response after primary HAV vaccination.
  Interventions: Drug: Vaqta Injectable Product

INTERVENTIONS:
Drug: Vaqta Injectable Product — Inactive vaccine against hepatitis A virus

SUMMARY:
Though HAV is mainly transmitted through the fecal-oral route, infection by sexual intercourse and blood transfusion is also possible. Injection drug users (IDUs) and men who have sex with men (MSM) have a higher risk of acquiring HAV due to their behaviors. Reemerging threat of hepatitis A among MSM in Taiwan has been reported recently. Based on the guidelines for the diagnosis and treatment of HIV/AIDS and the Advisory Committee on Immunization Practices (ACIP), Taiwan, vaccination of individuals against HAV with any of the following indications is recommended: HIV patients, adults with chronic hepatic disease, hemophilia, liver transplantation, occupational exposure, MSM, persons who use injection or noninjection illicit drugs, or persons traveling to or working in countries that have endemicity of HAV.

In HIV-infected patients, the immunogenicity to HAV vaccination is sub-optimal in HIV-infected patients and the seroconversion rate is estimated 68-90% after administration of 2 or 3 doses of HAV vaccine. Furthermore, the antibody titers of HIV-infected patients following HAV vaccination are significantly lower compared to those of HIV-uninfected persons. The sub-optimal response among HIV-infected subjects remains an unresolved problem. In this study, the investigators aim to determine the to conduct a randomized clinical trial to compare the immunogenicity of 2 different doses of HAV vaccination (1 dose versus 2 doses) in HIV-infected patients who failed to achieve serologic response in the primary vaccination. This proposal will provide the solid evidence to elucidate the role of booster HAV vaccination in HIV-infected patients without response to primary HAV vaccination.

DETAILED DESCRIPTION:
Though HAV is mainly transmitted through the fecal-oral route, infection by sexual intercourse and blood transfusion is also possible. Injection drug users (IDUs) and men who have sex with men (MSM) have a higher risk of acquiring HAV due to their behaviors. Acute hepatitis A outbreaks have been reported among these groups of patients in the USA, Europe and Australia. Reemerging threat of hepatitis A among MSM in Taiwan has been reported recently. HAV is generally a self-limited disease with marginal public health impact in countries with low HAV endemicity. HAV infection does not progress to chronic hepatitis and liver cirrhosis, but acute HAV infection poses a risk of acute liver failure or even death, particularly the persons with chronic HBV or HCV infection who develop super-infection with HAV.

In HIV-infected patients, liver disease is one of the three most common causes of death, and acute HAV infection is one cause of liver damage in HIV-infected patients. HIV-infected patients may experience prolonged HAV viremia, which can increase the risk of transmission to others. Furthermore, given that drug-induced liver injury associated with highly active antiretroviral therapy (HAART) and that HIV-infected subjects are frequently coinfected with HBV and HCV, these patients are considered especially susceptible to severe complications when they become infected by HAV. Risk factors for HIV infection, including MSM, IDUs, persons with multiple heterosexual contacts, and persons frequently exposed to blood and blood products, are also risk factors for HAV infection, since infection may occur through shared transmission routes. Based on the guidelines for the diagnosis and treatment of HIV/AIDS and the Advisory Committee on Immunization Practices (ACIP), Taiwan, vaccination of individuals against HAV with any of the following indications is recommended: HIV patients, adults with chronic hepatic disease, hemophilia, liver transplantation, occupational exposure, MSM, persons who use injection or noninjection illicit drugs, or persons traveling to or working in countries that have endemicity of HAV. The number of people living with HIV had grown to >28,000 persons by 2014 in Taiwan and MSM accounted for more than 50 % among all HIV-infected patients. Therefore, protection against HAV infection is essential in the care of HIV-infected patients.

The response rate to HAV vaccination is almost 100% among HIV-uninfected persons who receive 2 standard doses of HAV vaccine. However, the immunogenicity to HAV vaccination is sub-optimal in HIV-infected patients and the seroconversion rate is estimated 68-90% after administration of 2 or 3 doses of HAV vaccine. Furthermore, the antibody titers of HIV-infected patients following HAV vaccination are significantly lower compared to those of HIV-uninfected persons. Though one randomized clinical trial in HIV-infected patients suggested the 3-dose schedule of HAV vaccination tended to achieve a higher seroconversion rate than the 2-dose schedule at week 72 (78.3% versus 61.2%; P = 0.07), the optimal doses of HAV vaccine in these subjects remained unclear. Recently, the research group from National Taiwan University Hospital leaded by the principle investigator in this proposal published the findings in Hepatology that the serologic response rate to 2 and 3 doses of HAV vaccine was similar in HIV-infected MSM (75.7 % and 77.8 % seroconversion rate at week 48 for 2 doses and 3 doses, respectively). Administration of HAV vaccine in HIV-infected patients with higher CD4 counts (preferably >200 cells/μL) and suppression of HIV replication increased the seroconversion rate. This study provided the evidence that 2 doses of primary HAV vaccine was appropriate regimen in HIV-infected subjects. However, this study also found that the seroconversion rate (75.7 % and 77.8 % in 2 doses and 3 doses, respectively) in HIV-infected patients was lower than that in two-dose HIV-uninfected MSM (88.5 %). Around 20 patients receiving 2 doses of HAV vaccine and 30 patients with 3 doses of HAV vaccine did not have achieve seroconversion. This study based on Taiwanese population is the milestone for the research regarding HAV vaccination in HIV-infected patients. It not only demonstrates the safety of 2 or 3 doses of HAV vaccine among HIV-infected patients, but also gives as insight about the doses of primary vaccination. It is notable that the sub-optimal response among HIV-infected subjects remains an unresolved problem. The role of booster vaccination in HIV-infected patients without response to primary HAV vaccination has rarely been addressed in the literature. In one recent study conducted in Brazil, 23/29 (79.3%) from HIV-infected patients maintained HAV antibodies 7 years after primary HAV vaccination. The group that lost HAV seropositivity was revaccinated and 83.3% (5/6) responded with antibodies >20 mUI/mL after 2 doses of HAV vaccine. Though the limited numbers in this study, the data suggest that antibody titer monitoring is necessary in HIV-infected patients and revaccination is advisable to maintain protective levels of antibodies.

Although vaccination against HAV is essential for HIV-infected patients, the uptake of HAV vaccine is reported to be low. Studies of HAV vaccination coverage and screening rate for exposure to HAV in HIV patients are also limited. It is obvious that physicians interested in HIV care and vaccination planning is crucial to deal with this problem. In this study, we aim to determine the seroprevalence of HAV infection, the vaccine coverage rate and the factors associated with seropositivity in persons with HIV infection who sought HIV care over the past 6 years (2010-2016). Furthermore, the investigators aim to conduct a randomized clinical trial to compare the immunogenicity of 2 different doses of HAV vaccination (1 dose versus 2 doses) in HIV-infected patients who failed to achieve serologic response in the primary vaccination. This proposal will provide the solid evidence to elucidate the role of booster HAV vaccination in HIV-infected patients without response to primary HAV vaccination.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive individuals aged 20 year or more, and
* Those who had completed at least a primary series of HAV vaccination (i.e. two doses of HAVRIX 1440, 6-12 months apart; or two doses of Vaqta 50U, 6-18 months apart), and
* Those who failed to achieve serological response at least 4 weeks after the last dose of primary HAV vaccination.

Exclusion Criteria:

* Patients who have acute illness or acute hepatitis A related symptoms (fever, malaise, nausea, vomiting, abdominal discomfort, and jaundice) within 30 days.
* Patients who have positive anti-HAV IgM within 30 days.
* Patients who were taking immunosuppressant or steroid.
* Patients who were allergic to HAV vaccine.
* Incompetent or unconsented patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Serological responses at week 48 | Week 48
  Serological responses to HAV vaccination at week 48 after boosting vaccination

OTHER OUTCOMES:
Vaccine reaction | Vaccine reaction within 28 days after HAV vaccination
  Vaccine reaction after HAV vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Ching Hung, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen GJ, Sun HY, Lin KY, Hsieh SM, Chuang YC, Liu WD, Huang YS, Pan SC, Wu UI, Cheng A, Huang YC, Wu CH, Su YC, Liu WC, Chang SY, Hung CC. A Randomized Clinical Trial of 1-Dose vs Accelerated 2-Dose Schedule for Hepatitis A Virus (HAV) Revaccination Among People With Human Immunodeficiency Virus Who Were Nonresponders or Had Seroreversion After Primary HAV Vaccination. Clin Infect Dis. 2023 Aug 22;77(4):529-536. doi: 10.1093/cid/ciad206. PMID 37036404